CLINICAL TRIAL: NCT03788512
Title: Coexistence of Cerebral and Coronary Atherosclerosis in Acute Ischemic Cerebrovascular Disease Patients Registry
Acronym: CoCCA
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Xin Ma, Principal investigator, Xuanwu Hospital, Beijing
Other Study IDs: CoCCA
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Coexistence of Cerebral and Coronary Atherosclerosis; Acute Ischemic Cerebrovascular Disease
Keywords: acute ischemic cerebrovascular disease; cerebral atherosclerosis; coronary atherosclerosis; coexistence
MeSH Terms: conditions — Coronary Artery Disease; Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — anticoagulant peripheral blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AICVD patients with CoCCA: acute ischemic cerebrovascular disease patients with coexistence of cerebral and coronary atherosclerosis.
  Interventions: Other: observational only- no intervention

INTERVENTIONS:
Other: observational only- no intervention — observational only- no intervention

SUMMARY:
Coexistence of Cerebral and Coronary Atherosclerosis in Acute Ischemic Cerebrovascular Disease Patients Registry (CoCCA) is a single-center observational registry of patients hospitalized for acute ischemic cerebrovascular disease (AICVD) with atherosclerotic changes in both cerebral and coronary arteries.

This registry aims to establish quantified risk stratification and prognostic models, as well as suggest effective diagnostic and therapeutic strategies.

DETAILED DESCRIPTION:
Atherosclerosis has exerted huge global burden as the common pathological process underlying ischemic heart disease and cerebrovascular disease. A substantial portion of acute ischemic cerebrovascular disease (AICVD) patients have both cerebral and coronary atherosclerosis, which is an omen of poor outcomes. But there is large evidence gap in these high-risk patients' prognosis-related factors, limiting the improvement of care quality.

Coexistence of Cerebral and Coronary Atherosclerosis in Acute Ischemic Cerebrovascular Disease Patients Registry (CoCCA) is a single-center prospective observational registry of patients hospitalized for AICVD with atherosclerotic changes in both cerebral and coronary arteries.

This registry aims to establish quantified risk stratification and prognostic models, as well as suggest effective diagnostic and therapeutic strategies.

The clinical, imaging and laboratory information will be collected at the baseline. During an estimated 5-year follow-up, the vessel-related diagnostic or monitoring procedures, treatment, functional status and new vascular events will be recorded by web-based patients' self-reports, investigators' regular telephone visits.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as ischemic stroke or transient ischemic attack (TIA).
2. Less than 30 days after onset of ischemic stroke or TIA symptoms.
3. Extracranial or intracranial cerebral atherosclerosis confirmed by vascular ultrasound or CT angiograpgy or MR angiograpgy or digital substraction angiography.
4. Coronary atherosclerosis confirmed by CT angiograpgy or MR angiograpgy or digital substraction angiography; or with myocardial ischemia symptoms confirmed using electrocardiogram or echocardiography or cardiac MR; or with a history of percutaneous coronary intervention or coronary artery bypass graft.

Exclusion Criteria:

1. With malignant tumors or poor organ functions or hematologic diseases, whose estimated life expectancy is less than 5 years.
2. Patients refuse to participate in the research.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute ischemic cerebrovascular disease patients with coexistence of cerebral and coronary atherosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Cardiovascular Events | 1 year
  cardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death), ischemic stroke, myocardial infarction and unstable angina

SECONDARY OUTCOMES:
Rate of Major Adverse Cardiovascular Events | 90 days
  cardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death), ischemic stroke, myocardial infarction and unstable angina
Functional Outcome | 90 days
  Percentage of patients with modified Rankin Scale (mRS) scores (minimum 0 and maximum 5) 3 to 5, who are considered to be disabled.
Rate of Ischemic Stroke | 1 year
  fatal and nonfatal ischemic stroke.
Rate of Acute Coronary Syndrome | 1 year
  fatal and nonfatal myocardial infarction and unstable angina
Rate of Cardiovascular Mortality | 1 year
  any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death
Time to First Major Adverse Cardiovascular Event | 5 years
  from the date of enrollment until the date of first documented cardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death), ischemic stroke, myocardial infarction or unstable angina, whichever comes first, assessed up to 5 years
Time to First Ischemic Stroke | 5 years
  from the date of enrollment until the date of first documented ischemic stroke, assessed up to 5 years
Rate of Major Adverse Cardiovascular Events | 5 years
  cardiovascular mortality (any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death), ischemic stroke, myocardial infarction and unstable angina
Rate of Ischemic Stroke | 5 years
  fatal and nonfatal ischemic stroke
Rate of Acute Coronary Syndrome | 5 years
  fatal and nonfatal myocardial infarction and unstable angina
Rate of Cardiovascular Mortality | 5 years
  any mortality due to ischemic stroke, myocardial infarction, other cardiac diseases, or unobserved sudden death

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, BJ, China